CLINICAL TRIAL: NCT04597866
Title: Treatment of Complex Regional Pain Syndrome, a Qualitative Interview Study and a Case Series With Long-term Follow-up
Brief Title: Treatment of Complex Regional Pain Syndrome, a Long-term Follow-up
Acronym: TORNADO
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-03383
Record Dates: First submitted 2020-09-15; First posted 2020-10-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Complex Regional Pain Syndromes; Chronic Pain
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRPS
  Interventions: Behavioral: Multimodal rehabilitation

INTERVENTIONS:
Behavioral: Multimodal rehabilitation — A combination of exposure in vivo and interventions directly targeting the cortical reorganization for treating CRPS.

SUMMARY:
Complex regional pain syndrome, CRPS, is an uncommon but often very disabling chronic pain syndrome characterized by, beside pain: sensory disturbances, peripheral autonomic changes and inflammatory features. The diagnosis is subdivided in CRPS type 1 where no nerve injury has been identified, and CRPS type 2 when a major nerve injury has been verified.

A combination of exposure in vivo, a form of behaviour therapy where the patient is gradually confronted with avoided movements and activities, and interventions directly targeting a hypothesized cortical reorganisation is an interesting novel approach for treating CRPS.

The present study consists of (1) a qualitative interview study with 10-15 subjects that has received this form of treatment, in order to better understand their experience and effects of the treatment, and (2) a case series with long-term follow-up of 3-5 subjects that received the treatment för 5-8 years ago, in order to study the long term effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has participated in multimodal treatment for CRPS at Uppsala University Hospital

Exclusion Criteria:

* Other serious physical or mental condition

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with CRPS 1 or 2, diagnosed according to the Budapest criteria that has received in-patient treatment at Uppsala University Hospital, comprised of graded exposure therapy in vivo, in combination with methods targeting cortical reorganisation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis | 1 day
  Whether the subject still fulfill diagnostic criteria for CRPS
Subjective experience | 1 day
  A qualitative interview targeting the subjects own experience of the treatment and its effect

SECONDARY OUTCOMES:
Level of pain | 1 day
  Subjective level of pain on a Likert-scale 0-10 (NRS)
Subjective experience of quality of life | 1 day
  Quality of life, measured with the RAND-36 (0-100, higher scores mean a better outcome)
Global impression of change | 1 day
  Global impression of change measured with a single question (0-6, higher scores mean a better outcome)
Acceptance of pain | 1 day (0-156, higher scores mean a better outcome)
  Measured with the Chronic Pain Acceptance Questionnaire, CPAQ (0-156, higher scores mean a better outcome)
Fear of pain | 1 day (0-52, lower scores mean a better outcome)
  Measured with the Tampa Scale of Kinesiophobia, TSK (0-52, lower scores mean a better outcome)
Pain catastrophizing | 1 day (0-52, lower scores mean a better outcome)
  Measured with Pain Catastrophizing Scale, PCS (0-52, lower scores mean a better outcome)
Avoidance of activities | 1 day (0-100, lower scores mean a better outcome)
  Measured with the Photograph Series of Daily Activities, PHODA (0-100, lower scores mean a better outcome)
Neglect of the affected limb | 1 day (0-36, lower scores mean a better outcome)
  Measured with a five item questionnaire (0-36, lower scores mean a better outcome)
Subjective experience of quality of life 2 | 1 day
  EuroQol 5D, EQ-5D (0-15, higher scores means a better outcome)
Subjective experience of quality of life 3 | 1 day
  Life Satisfaction Questionnaire, LiSat 11 (11-66, higher scores means a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Bothelius, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided